CLINICAL TRIAL: NCT05360303
Title: Interest of Electroneuromyography in the Diagnosis of Thoracic Outlet Syndrome
Brief Title: Electromyography in Thoracic Outlet Syndrome
Acronym: ENMG-AFC
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC22_0229
Record Dates: First submitted 2022-04-25; First posted 2022-05-04 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Thoracic Outlet Syndrome
Keywords: Thoracic outlet syndrome; electromyography; neurogenic; rehabilitation; diagnosis
MeSH Terms: conditions — Thoracic Outlet Syndrome; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trial population: No Intervention but evaluation of the electroneuromyography at the M1 visit for patients with a clinical diagnostic of thoracic outlet syndrome.

SUMMARY:
Record the ENMG data carried out systematically in patients treated by rehabilitation for thoracic outlet syndrome in order to assess their characteristics and judge the relevance of these data in the context of the diagnosis and their possible modifications following the rehabilitation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient rehabilitation for thoracic outlet syndrome
* Patients' agreement

Exclusion Criteria:

* < 18 years old
* Not able to consent
* Pregnancy
* Musculoskeletal disorders of the upper limbs
* Acute cardiac, pulmonary, metabolic or neurological diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a thoracic outlet syndrome who will be included during their usual rehabilitation management. They will benefit from the usual Electromyography of stimulodetection with surface electrodes at the beginning of the management. The same examination will be performed at the end of the treatment to evaluate the impact of the rehabilitation on the electrophysiological results and to orientate, if necessary, towards a potential surgery.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-03-23 (Actual)

PRIMARY OUTCOMES:
Evaluation of the presence of ENMG abnormality and in particular on the medial cutaneous nerve of the forearm of patients with a clinical diagnosis of TOS | 0 Month
  Conduction abnormality of the medial cutaneous nerve of the forearm

SECONDARY OUTCOMES:
Evaluation of ENMG changes following rehabilitation treatment of patients | 1 Month
  evolution of electrophysiological changes following treatment
Evaluation of ENMG changes following rehabilitation treatment of patients | 1 Month
  evolution of the Visual Analog Score for pain (scale from 0 to 10 ; 10 being the worst outcome)
Evaluation of ENMG changes following rehabilitation treatment of patients | 1 Month
  evolution of the Quick Disabilities of the Arm, Shoulder and Hand Score (scale from 0 to 100 ; 100 being the worst outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Medicine and Locomotive Rehabilitation (Nantes University Hospital), Nantes, France

IPD SHARING:
Plan to Share IPD: No